CLINICAL TRIAL: NCT04953936
Title: β-hydroxy-β-methylbutyrate-enriched Nutritional Supplements for Obesity Adults During Weight Loss: a Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: β-hydroxy-β-methylbutyrate-enriched Nutritional Supplements for Obesity Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yuxiang Liang, Physiotherapist, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021（202）
Record Dates: First submitted 2021-06-12; First posted 2021-07-08 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMB (Experimental): The participants will receive oral HMB-enriched nutritional supplements (65 g once daily)
  Interventions: Dietary Supplement: HMB-enriched Nutritional Supplements; Behavioral: Caloric Restrition Diet
- Placebo (Placebo Comparator): The participants will receive a placebo (maltodextrin 65 g once daily) with the same package as the intervention.
  Interventions: Dietary Supplement: Placebo; Behavioral: Caloric Restrition Diet

INTERVENTIONS:
Dietary Supplement: HMB-enriched Nutritional Supplements — The participants will receive oral HMB-enriched nutritional supplements (65 g, once daily), which include soybean isolate protein, flaxseed oil powder, yam powder, whey protein, oligomeric isomaltose powder, cocoa powder, medium-chain fatty acid powder, calcium beta-hydroxy-beta-methylbutyrate, sunflower seed oil powder, L-glutamine, wheat germ powder, membrane isolated casein, wheat oligopeptide, konjac flour, vitamin E, vitamin D, stevioside, edible flavors.
  Arms: HMB
Dietary Supplement: Placebo — Placebo (maltodextrin 65 g once daily) with the same package as the intervention.
  Arms: Placebo
Behavioral: Caloric Restrition Diet — Caloric restriction diet with individualized nutritional guidance from professional dietitians by video regarding caloric restriction strategies

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of HMB-enriched nutritional supplements for improving muscle mass and muscle function in Chinese adults with obesity during the weight loss process using calorie restriction.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 30-50 years
2. Currently having obesity defined by body mass index (BMI) ≥ 28 kg/m2 (based on measured body weight and height at booking, using validated scales)
3. Having an intention to lost weight via caloric restriction
4. Apparently healthy and able to walk independently
5. Able to eat independently to meet their energy needs
6. Without significant body weight change in the last 6 month (less than 5% change in body weight)
7. Having sedentary habit defined by Sedentary Behavior Research Network
8. Able to collaborate with the research staff.

Exclusion Criteria:

1. Having a history of intolerance to enteral nutrition, food (e.g., lactose intolerance), or being allergic to the components of our HMB-enriched nutritional supplements (e.g., soy or corn);
2. Having any implants (e.g., pacemakers);
3. Current use of other nutritional supplements or drugs that may have an impact on the effectiveness of the intervention (e.g., glucocorticoids, antineoplastic drugs, antituberculosis drugs, sedatives, antipsychotics, muscle relaxants, monoamine oxidase inhibitors, antibiotics) within 3 months prior to enrollment;
4. Secondary obesity caused by diseases (e.g., hypothalamic diseases and hypercortisolism) or drugs (e.g. glucocorticoids, insulin, tricyclic antidepressants);
5. Clinically visible edema;
6. Trauma, surgery, hospitalization, fall, or fracture within 6 months prior to enrollment;
7. Pregnancy, having pregnancy plans, or lactation;
8. Individuals who are participating in other clinical trials; any acute illness (e.g., acute infection, myocardial infarction, arrhythmia, myocarditis, appendicitis, etc.);
9. Swallowing disorders; abnormal thyroid function (including hyperthyroidism and hypothyroidism);
10. Having a history of diabetes, respiratory diseases, cardiovascular diseases, uncontrolled hypertension, kidney diseases, digestive system diseases, renal insufficiency, mental illness, neurological diseases, hematologic diseases, liver diseases (except for fatty liver), chronic infection (e.g., tuberculosis), immune system diseases, joint disorders, any type of tumor;
11. Alcohol consumption over two standard alcoholic beverages (20 g of alcohol/day);
12. Difficulty to comply with the study protocol;
13. Other conditions that indicate the individuals are inappropriate for participation in this study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean change in whole-body skeletal muscle mass (SMM) | 12 weeks
  The whole-body skeletal muscle mass (SMM)

SECONDARY OUTCOMES:
The mean change in appendicular skeletal muscle mass (ASMM) | 12 weeks
  These data will be measured using InBody 770 (Biospace Co., Seoul, Korea).
The mean change in trunk skeletal muscle mass (TSMM) | 12 weeks
  These data will be measured using InBody 770 (Biospace Co., Seoul, Korea).
The mean change in total body fat mass (BFM) | 12 weeks
  These data will be measured using InBody 770 (Biospace Co., Seoul, Korea).
The mean change in total appendicular body fat mass (ABFM) | 12 weeks
  These data will be measured using InBody 770 (Biospace Co., Seoul, Korea).
The mean change in trunk body fat mass (TBFM) | 12 weeks
  These data will be measured using InBody 770 (Biospace Co., Seoul, Korea).
The mean change in basal metabolic rate (BMR) | 12 weeks
  These data will be measured using InBody 770 (Biospace Co., Seoul, Korea).
The mean change in phase angle (PA) | 12 weeks
  These data will be measured using InBody 770 (Biospace Co., Seoul, Korea).
The mean change in body weight (BW) | 12 weeks
  These data will be measured using InBody 770 (Biospace Co., Seoul, Korea).
The mean change in handgrip strength (HGS) | 6 and 12 weeks
  A trained nurse will measure HGS using a digital handheld dynamometer (EH101; Xiangshan Inc, Guangdong, China) to the nearest 0.1 kg .
The mean change in waist circumference | 6 and 12 weeks
  A trained nurse will measure waist circumference using a tape at the level midway between the lower rib margin and the iliac crest with the participant breathing out gently.
The mean change in hip circumference | 6 and 12 weeks
  Hip circumference was measured as the maximum circumference over the buttocks
The mean change in physical activity | From the beginning to weeks 3, 6, 9, and 12.
  It will be measured using self-reported International Physical Activity Questionnaire Short Form (IPAQ-SF).The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires. Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health related physical activity.
The mean change in the score of the sit-to-stand test | 6 and 12 weeks
  A trained nurse will perform the 30-second sit-to-stand test ,which is a classic test for measuring the performance of lower extremity muscles.
The mean change in energy intake | From the beginning to weeks 3, 6, 9, and 12
  It will be measured for all participants using the self-reported Food Frequency Questionnaire (FFQ)
The mean change in lipid profiles | 12 weeks
  It will be tested using standard method.
The mean change in fasting glucose | 12 weeks
  It will be tested using standard method.
The mean change in fasting insulin | 12 weeks
  It will be tested using standard method.
The mean change in HOMA-IR | 12 weeks
  It will be tested using standard method.
The mean change in albumin | 12 weeks
  It will be tested using standard method.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Yang, Study Chair — West China Hospital; Jiaojiao Jiang, Study Director — West China Hospital
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jing X, Liang Y, Wang R, Fu H, Jiang J, Yang M. beta-hydroxy-beta-methylbutyrate-enriched nutritional supplements for obese adults during weight loss: study protocol of a randomised, double-blind, placebo-controlled clinical trial. BMJ Open. 2022 Jun 23;12(6):e055420. doi: 10.1136/bmjopen-2021-055420. PMID 35738656